CLINICAL TRIAL: NCT07404826
Title: A Randomized, Sham Controlled Clinical Trial to Assess the Effectiveness of a Positive End Expiratory Device for Accelerating and Maintaining Pulmonary Rehabilitation Gains
Brief Title: PEP Buddy in Pulmonary Rehabilitation
Acronym: PEPR
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRD6-010-24W; 1I01RD000440-01A2 (Other Grant/Funding Number: VA ORD); 25-81 (Other: VA Central IRB Proposal Number)
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: COPD
Keywords: Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants will be block randomized in groups of varying sizes to either PEP Buddy or sham. The PEP Buddy and sham groups will run in parallel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and research team will be blinded. Participants will be provided with a device in an opaque box, both PEP Buddy and sham packaging will be the same. The dives themselves will look similar and the difference between PEP Buddy and sham will not be able to be determined by the naked eye.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PEP Buddy (Experimental): This arm will be provided with a portable device that provides 5-7 cm H2O of expiratory pressure, to be used when subjectively breathless
  Interventions: Device: PEP Buddy
- Sham (Sham Comparator): This arm will be provided with a portable device that appears the same as PEP Buddy but provides 1-3 cm H2O of expiratory pressure, to be used when subjectively breathless
  Interventions: Device: PEP Buddy Sham

INTERVENTIONS:
Device: PEP Buddy — This is a small, portable device worn about the neck with a lanyard, that can be used to control symptoms of breathlessness associated with chronic lung disease.
  Arms: PEP Buddy
Device: PEP Buddy Sham — A Device that appears the same as PEP Buddy but only provides the expiratory pressure of the standard-of-care pursed lip breathing
  Other Names: Sham
  Arms: Sham

SUMMARY:
In this study, the investigators will test Veterans with COPD in Pulmonary Rehabilitation. Between two groups, the investigators will give one group a device that assists with breathing and symptoms and the other receives a 'sham' device which does not provide these benefits. The investigators will test to see if the symptoms and exercise capacity of the group who receives this device improves faster in Pulmonary Rehabilitation and has longer lasting benefits after the end of Pulmonary Rehabilitation.

DETAILED DESCRIPTION:
In this randomized, double-blinded, sham-controlled clinical trial, the investigators will test the effectiveness of the use of a positive expiratory device (PEP Buddy) vs. sham in participants with COPD in Pulmonary Rehabilitation and after discharge from Pulmonary Rehabilitation for up to one year. The investigators will compare changes in quality of life metrics and measurements of functional capacity between the intervention and sham groups over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Referral to Pulmonary Rehabilitation for COPD
* FEV1 <80% predicted
* Participants must be able to exercise on 4L/m nasal cannula O2

Exclusion Criteria:

* Those deemed by the study personnel to have a lung disease other than COPD impacting their daily dyspnea
* Those that are unable to perform study procedures or are unwilling or unable to use PEP Buddy
* Those that have a component of lung disease driven by aspiration or neurological conditions affecting the face or oropharynx
* Those with a life expectancy of <1 year
* Those with a known surgical intervention that will require a prolonged recovery in the year after enrollment
* Those with a malignancy beyond Stage I or non-melanoma skin cancer
* Those shown shown to have memory loss of MOCA testing

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-03-29 (Estimated); Study Completion 2030-03-29 (Estimated)

PRIMARY OUTCOMES:
San Diego Shortness of breath Questionnaire | 12 Months
  This is a standardized survey used to quantify the impact of daily respiratory symptoms on quality of life. This will be collected on enrollment and the investigators will compare the change between groups at Weeks 3, 6, 9, and 12 and at six-and twelve-months after enrollment.
Daily steps measured by wrist-wron accelerometer | 12 Months
  Using accelerometry, the investigators will show the changes in daily step counts between groups over the one year of time in the study.

SECONDARY OUTCOMES:
One-Minute Sit to Stand test | 12 Months
  The investigators will perform this test at enrollment and at weeks 3, 6, 9, and 12 as well as six-and twelve-months after enrollment and compare between groups. This test calculates the number of times a participant can sit and rise from a chair over the course of a minute.
Six Minute Walk Test | 12 months
  A standard test of exercise capacity in those with chronic lung disease. The investigators will assess changes in the six-minute walk test difference from enrollment at Weeks 3, 6, 9, and 12 in the study and at six-and twelve-months after the conclusion of the study.
St. George Respiratory Questionaire | 12 Months
  The investigators will compare the values between groups from enrollment at Weeks 3, 6, 9, and 12 and at six-and twelve-months after enrollment. This is a standard survey form in which participants report the severity and daily impact of respiratory symptoms and how they may inhibit daily activity.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Matthew Burkes, MD MS, Principal Investigator — Cincinnati VA Medical Center, Cincinnati, OH
Locations (2):
- United States (2):
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share data with VA researchers that will be de-identified via Safe Harbor approach. However, if a non-VA researcher requests aggregate data, the investigators will work with local research office, facility privacy officer, and information security officer to identify an applicable agreement for data sharing. No VA data will include any PHI to any non-VA researchers requesting VA data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will not be shared until the close of the study (March 2025). The investigators will then share data for six years after close of study.
Access Criteria: The investigators ask that any requesting entity contact the Primary Investigator by e-mail to begin a request for data via VA processes.